CLINICAL TRIAL: NCT06270758
Title: Clinical Validation of BBCT-hip Methodology for Femur Fracture Risk Prediction
Brief Title: Clinical Validation of BBCT-hip
Acronym: ValidaBBCT-hip
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 453/2023/Sper/IOR
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Osteoporosis
Keywords: hip fracture; fracture prediction; finite element; in silico; osteoporotic fracture
MeSH Terms: conditions — Osteoporosis; Hip Fractures; Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fractured subjects: Post-menopausal women who have been hospitalised because of a femur fracture.
  Interventions: Diagnostic Test: CT scan at the femur
- Control subjetcs: Post-menopausal women without history of fracture
  Interventions: Diagnostic Test: CT scan at the femur

INTERVENTIONS:
Diagnostic Test: CT scan at the femur — Additional CT scan which is not part of the standard clinical path

SUMMARY:
The clinical study is aimed at assessing the accuracy of the in silico methodology BBCT-hip. BBCT-hip takes as inputs the subject-specific height and weight, and the CT scan of his femur to predict the risk of fracture for the femur upon falling. In the study, 150 subjects who suffered from a fracture will be enrolled, in addition to 150 control subjects. CT scans will be carried out for both groups (no later than 3 months for the fracture group) and BBCT-hip run,in order that the risk of fracture will be obtained. First, a transversal study will be performed, where the stratification accuracy of BBCT-hip will be assessed in terms of the ability of the predicted risk of fracture to separate fracture and control subjects. Furthermore, the control subjets will be followed up to assess BBCT-hip predictive accuracy through a longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* caucasic post-menopausal women resident in Emilia-Romagna
* menopause (>= 45 years)

Exclusion Criteria:

* tumours
* not free living
* Chronic diseases with severe organ failure / endocrine diseases of parathyroid, thyroid, adrenal gland / intestinal malabsorption, osteomalacia / Paget bone / rheumatoid arthritis. Neurodegenerative diseases
* Long-term continuous therapy (>3 months) with corticosteroids and proton pump inhibitors or aromatase inhibitors
* Previous femur fractures
* Presence of hip/knee prosthesis

only for the fracturegroup:

* presence of fixation devices after the fracture
* femur fracture due to high energy trauma

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Study Population: Resident in Emilia Romagna, Italy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2030-11-06 (Estimated); Study Completion 2030-11-06 (Estimated)

PRIMARY OUTCOMES:
Femoral fracture event | 5 years
BBCT-hip risk prediction | 5 years

SECONDARY OUTCOMES:
T-score | 5 years
  gold standard parameter for osteoporosis diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Publication about BBCT-hip methodology — https://link.springer.com/article/10.1007/s10439-022-02924-1